CLINICAL TRIAL: NCT04251182
Title: A Randomized, Double-Blind, Placebo-Controlled Multi-Center Study to Evaluate the Safety and Efficacy of Three Dose Strengths of T3D-959 in Subjects With Mild-to-Moderate Alzheimer's Disease
Brief Title: Clinical Study Evaluating Efficacy and Safety of T3D-959 in Mild-to-moderate AD Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: T3D Therapeutics, Inc. (Industry)
Collaborators: National Institute on Aging (NIA) (NIH); Clinilabs, Inc. (Other); Alzheimer's Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: T3D959-202; 1R01AG061122 (NIH)
Record Dates: First submitted 2020-01-24; First posted 2020-01-31 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Alzheimer Disease
Keywords: mild-to-moderate Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, placebo-controlled design evaluating three dose levels (15 mg, 30 mg, 45 mg) of T3D-959 in subjects with mild-to-moderate Alzheimer's Disease. Subjects will be stratified by ApoE4 genotype and assigned to one of four dose groups (1:1:1:1 ratio) in a randomized fashion.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study drug packaging and labeling will maintain the double-blind design of the study. T3D-959 and placebo capsules will be identical in appearance. Therefore, the subject's treatment assignment will not be known to the subject or the study site personnel. None of the persons directly involved in the conduct of the study will have access to the treatment code. The DSMB and persons involved with reporting to the DSMB (as outlined within the DSMB Charter) will have access to the treatment code. The treatment code will be released to the study team after the study database has been locked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo, matching T3D-959 active capsules, is pregelatinized starch NF, magnesium stearate NF, and size 0, hard gelatin, white/white, opaque, unmarked capsules. Subjects randomized to placebo will ingest three size 0 placebo capsules once per day in the morning.
  Interventions: Drug: Placebos
- 15mg T3D-959 (Experimental): T3D-959 15 mg dose: T3D-959 is a small molecule dual nuclear receptor agonist that regulates transcription of genes, in particular those involved in glucose energy and lipid metabolism. T3D-959 is 15-times more potent for PPAR delta than for the secondary target of the drug, PPAR gamma. The 15 mg strength contains 15mg T3D-959, pregelatinized starch NF, magnesium stearate NF, and size 0, hard gelatin, white/white, opaque, unmarked capsules. Subjects will ingest one size 0, 15mg capsule and two placebo capsules once per day in the morning.
  Interventions: Drug: 15mg T3D-959
- 30mg T3D-959 (Experimental): T3D-959 30 mg dose: Subjects will ingest two size 0, 15mg capsules and one placebo capsule once per day in the morning.
  Interventions: Drug: 30 mg T3D-959
- 45mg T3D-959 (Experimental): T3D-959 45 mg dose: Subjects will ingest three size 0, 15mg capsules once per day in the morning.
  Interventions: Drug: 45 mg T3D-959

INTERVENTIONS:
Drug: 15mg T3D-959 — Oral administration once daily in the morning
  Other Names: T3D-959
  Arms: 15mg T3D-959
Drug: 30 mg T3D-959 — Oral administration once daily in the morning
  Other Names: T3D-959
  Arms: 30mg T3D-959
Drug: 45 mg T3D-959 — Oral administration once daily in the morning
  Other Names: T3D-959
  Arms: 45mg T3D-959
Drug: Placebos — Oral administration once daily in the morning
  Other Names: T3D-959 Placebo
  Arms: Placebo

SUMMARY:
A Randomized, Double-Blind, Placebo-Controlled Multi-Center Study to Evaluate the Safety and Efficacy of Three Dose Strengths of T3D-959 in Subjects with Mild-to-Moderate Alzheimer's Disease.

DETAILED DESCRIPTION:
Study Design & Methods: Phase 2 multi-center, randomized, double blind, placebo-controlled study of T3D959 15 mg, 30 mg, 45 mg, or matching placebo administered orally once daily for 24 weeks. There will be equal allocation of subject numbers across the four groups. Stratified randomization will be conducted on the basis of ApoE4 genotype so that subjects are randomized into one of the four dose groups within each stratum of ApoE4 status: ApoE4-positive (at least one E4 allele) vs ApoE4-negative (no E4 alleles).

Following informed consent, subjects will enter the screening phase of the study.

Once eligibility is confirmed and before the start of the first dose of study drug, subjects will be randomized on a 1:1:1:1 basis to placebo or T3D959 treatment (15mg, 30mg, 45mg) for the 24-week treatment period. Investigators, subjects, and caregivers will be blinded to the treatment assignment.

Study schedule visits: screening, baseline, weeks 4, 8, 16, 24 and 28 (F/U visit)

ELIGIBILITY:
Inclusion Criteria:

* Have a reliable caregiver, an identified adult who, in the opinion of the investigator has sufficient contact to knowledgeably report on the subject's daily cognition, function, behavior, safety, compliance and adherence. Same caregiver(s) must assist the subject throughout the duration of the trial.
* Have a clinical diagnosis of mild-to-moderate AD (Stage 4 or 5) according to the NIA-AA (National Institute of Aging - Alzheimer's Association) criteria at screening
* Meet criteria for mild-to-moderate cognitive impairment with Mini-Mental State Examination (MMSE) score of 14 through 26 at the screening visit.
* Neuroimaging evidence consistent with the diagnosis of AD
* Modified Hachinski </= 4 at screening
* Clinical Dementia Rating is 0.5 to 2.0 at screening and Clinical Dementia Rating - Sum of Boxes is ≥ 3 at screening
* Visual and auditory acuity adequate for neuropsychological testing
* No evidence of hepatic impairment or renal insufficiency

Exclusion Criteria:

* Have a current diagnosis of a significant psychiatric illness per the Diagnostic and Statistical Manual of Mental Disorders V (DSM-V)
* With untreated clinical depression (GDS >/= 6 at screening and baseline)
* Have a current diagnosis of a neurological disease other than AD
* With glycosylated hemoglobin (HbA1c) >/= 7.7 at screening
* With a diagnosis of unstable diabetes
* With clinically significant thyroid disease at screening TSH >5
* Have any of the following values at the screening visit:

  * ALT and/or AST value that is twice the upper limit of normal
  * Total bilirubin value that exceeds 2 mg/dL
  * Creatinine level >1.5 mg/dL in men or > 1.4 mg/dL in women
  * Positive urinalysis (other than trace result) unless a cause other than renal impairment
  * Glomerular filtration rate (GFR) values <54 mL/min/1.73 m2
  * Gamma-glutamyl transpeptidase (GGT) value that is twice the upper limit of normal
  * Is positive for hepatitis B or anti-hepatitis C virus antibodies at the screening
* Have a history of moderate or severe congestive heart failure, NYHA class III or IV
* Have experienced a previous cardiovascular event (myocardial infarct, by-pass surgery, or PTCA) within the past 12 months prior to the baseline
* Have blood pressure reading at screening that is greater than 160/100 mmHg
* Have a clinically significant unstable illness
* Have a history of HIV infection
* Have a history of alcohol, drug abuse or dependence
* Have a history of cancer within 5 years of the screening
* Have any surgical or medical condition which may significantly alter the absorption of any drug substance
* Females who are pregnant, nursing or of childbearing potential and not practicing effective contraception
* Is required to take excluded medications as specified protocol
* Have a known or suspected intolerance or hypersensitivity to the study drug, closely related compounds
* Resides in hospital or moderate to high dependency continuous care facility
* Are non-ambulatory, or wheelchair-bound
* Have evidence of clinically relevant pathology that in the investigator's opinion could interfere with the study results or put the subject's safety at risk
* History of swallowing difficulties

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-02-17 (Actual)

PRIMARY OUTCOMES:
Efficacy of T3D-959 on cognition | 28 weeks (Subjects are on active treatment for 24 weeks followed by a 4-week follow-up)
  Change in cognition as assessed by The Alzheimer's Disease Assessment Scale 11-task cognitive subscale (ADAS-Cog11) from baseline to end of treatment visit, compared to placebo
Efficacy of T3D-959 on function | 28 weeks (Subjects are on active treatment for 24 weeks followed by a 4-week follow-up)
  Change in global function as assessed by Alzheimer's Disease Cooperative Study Clinical Global Impression of Change (ADCS-CGIC) from baseline to end of treatment visit, compared to placebo
Safety and tolerability of T3D-959 | 28 weeks (Subjects are on active treatment for 24 weeks followed by a 4-week follow-up)
  Safety will be assessed by 1) AEs, clinical labs, ECG, weight, vital signs 2) Geriatric Depression Scale (GDS) 3)Columbia Suicide Severity Rating Scale (C-SSRS)

SECONDARY OUTCOMES:
Efficacy of T3D-959 on executive function | 28 weeks (Subjects are on active treatment for 24 weeks followed by a 4-week follow-up)
  Change in executive function as assessed by the Digit Symbol Coding Test (DSCT) from baseline to end of treatment visit, compared to placebo
Efficacy of T3D-959 on plasma Aβ 42/40 ratio biomarker level | 28 weeks (Subjects are on active treatment for 24 weeks followed by a 4-week follow-up)
  Change in Aβ 42/40 ratio plasma biomarker from baseline to end of treatment visit, compared to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Blake Swearingen, MS, Study Director — T3D Therapeutics, Inc.
Locations (1):
- T3D Therapeutics, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
A Clinical Study Report (CSR) will be generated within 9 months after database lock. Aggregate study data will be made available in this report.